CLINICAL TRIAL: NCT05450861
Title: Effect of the Composition From Fish on Promoting Hair Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KMUHIRB-F(I)-20190142
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Hair Loss/Baldness; Androgenic Alopecia; Male Pattern Baldness; Female Pattern Alopecia
Keywords: Hair Loss/Baldness; Androgenic Alopecia; male pattern baldness; female pattern alopecia; sfDNA
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant
Masking Description: using scalp conditioning solution without target composition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SF DNA Treatment (Experimental): the scalp conditioning solution with SF DNA extraction composition is applied daily and combination with hair loss medical treatment for eight weeks.
  Interventions: Other: SF DNA extraction composition
- Placebo (Placebo Comparator): the scalp conditioning solution without SF DNA extraction composition is applied daily and combination with hair loss medical treatment for eight weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: SF DNA extraction composition — the composition of small fragments of DNA from fish
  Arms: SF DNA Treatment
Other: Placebo — the scalp conditioning solution without SF DNA extraction composition
  Arms: Placebo

SUMMARY:
According to the World Health Organization data, one out of every five Chinese men has a hair loss symptom, and the hair loss is as high as 84% before the age of 30. Based on the experience of clinicians, there seems to be an increasing trend of alopecia patients who seek the treatment in Taiwan.

Treating pathological hair loss requires prompt diagnosis and management to prevent conditions that could lead to permanent hair loss. The current methods of treating hair loss include oral drugs, topical medication, laser illuminating treatment, platelet-rich plasma and hair transplant surgery. However, these treatments also have different disadvantages. Prolonged continuous use of oral and topical medications may be accompanied by side effects. Other treatment modalities may require higher costs, require return visits, or be more invasive.

Previous study found that the composition of small DNA fragments (SF DNA) possesses not only toxin-free in primary human skin cells and nude mice, but also inhibits inflammation and ROS generation in the process of skin aging. SF DNA also contributes to promote the proliferation and differentiation of hair follicles, and stimulates the hair growth in nude mice through affecting JAK-STAT pathway.

The investigators hypothesize that the clinical application of SF DNA scalp conditioning solution attenuates inflammatory responses, promotes the proliferation and differentiation of hair follicles, and increases the hair of hair loss patients and inspires the quality of life.

DETAILED DESCRIPTION:
Thick and healthy hair is a symbol, representing the attractiveness, youth, health and fertility of adults. However, according to the World Health Organization data, one out of every five Chinese men has a hair loss symptom, and the hair loss is as high as 84% before the age of 30. Based on the experience of clinicians, there seems to be an increasing trend of alopecia patients who seek the treatment in Taiwan.

Excessive hair shedding potentially distributes to physiological effect which is in the senile hair-loss/postpartum state, or pathological effect which is due to thyroid disturbances, trauma, lupus erythematosus, scleroderma, drug effects, iron deficiency, or fungal infection. There are also two kinds of pathological hair loss, alopecia areata and androgen-derived hair loss, both of them are difficult to treatment in clinical so far.

First-line interventions for treating excessive hair shedding include lifestyle modification and behavior therapy, such as clean scalp, adjusted daily routine, and alleviated psychological stress. The second-line interventions is drug therapy which is helpful in the treatment of excessive hair shedding, but respond to conservative measures. The minoxidil application is an effective treatment for androgenetic alopecia in both men and women. Its side effects include redness and scaling of the scalp. The finasteride reduces the dihydrotestosterone (DHT) in the serum and scalp, but it may cause sexual dysfunction. However, laser illuminating treatment, platelet-rich plasma (PRP) treatment, and surgical (hair transplant surgery) are cataloged to third-line interventions. The PRP treatment is safe, rapid, and process tolerable, and has the advantage of being finer and relatively low-cost compared to hair transplantation.

Follicular units pre-treatment by PRP also facilitate increase of the survival rate of transplanted hair. Although light therapy does not have the side effects of percutaneous or oral administration, treatment with two to three times a week can also cause problems for patients. Autologous hair transplantation is a supplementary treatment for advanced androgenetic alopecia. However, the cost of hair transplantation is high, and the survival rate of hair after transplantation is also worrying. In addition, surgery during convalescence also produces the costs of hospitalization and the loss of productivity. These problems are worthwhile for most patients with excessive hair shedding. To minimize invasiveness treatment, the efficacy, safety, and cost-effectiveness should be considered.

Our previous study found that the composition of small DNA fragments (SF DNA) possesses not only toxin-free in primary human skin cells and nude mice, but also inhibits inflammation and ROS generation in the process of skin aging. SF DNA also contributes to promote the proliferation and differentiation of hair follicles, and stimulates the hair growth in nude mice through affecting JAK-STAT pathway.

The investigators hypothesize that the clinical application of SF DNA scalp conditioning solution attenuates inflammatory responses, promotes the proliferation and differentiation of hair follicles, and increases the hair of hair loss patients and inspires the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 20~75 years old.
* Diagnosed with alopecia by dermatologists.
* Willing to maintain the same hair style, color, shampoo and hair products used, and approximate hair length starting from signing ICF and throughout the study.
* The subject can understand and obey order.

Exclusion Criteria:

* Pregnant, nursing, or planning a pregnancy during the study.
* Use of any topical medication (such as minoxidil or any other solution for hair growth), laser therapy, or chemotherapy, within the preceding 4 weeks.
* Personal medical history of abnormal blood clotting such as bleeding disorders or platelet dysfunction syndrome.
* Personal medical history of unstable vital signs such as hypotension or uncontrolled hypertension syndrome.
* Prior hair transplant.
* Chronic scalp disorders that require medications.
* Uses medication known to cause hair thinning such as Coumadin and anti- depressants/anti-psychotics.
* Existing scalp diseases such as folliculitis, scalp psoriasis, seborrheic dermatitis, or inflammatory scalp conditions.
* Enrolled in any other medical study or has been enrolled in any medical study in the past 6 months.
* Any hematologic abnormalities.
* Severe allergies manifested by a history of anaphylaxis, or history or presence of multiple severe allergies.
* Planned upcoming surgeries.
* Tattoo on scalp.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
hair density | 8 weeks
  using the hair scalp analysis device to measure hair density at the vertex baldness site.
hair diameter | 8 weeks
  using the hair scalp analysis device to measure hair diameter at the vertex baldness site.

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI) questionnaire | 8 weeks
  Participants answered the DLQI questionnaire by self. Higher scores mean a worse outcome (poor quality of life).

OTHER OUTCOMES:
hair density | 4 weeks
  using the hair scalp analysis device to measure hair density at the vertex baldness site.
hair diameter | 4 weeks
  using the hair scalp analysis device to measure hair diameter at the vertex baldness site.
DLQI questionnaire | 4 weeks
  Participants answered the DLQI questionnaire by self. Higher scores mean a worse outcome (poor quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Municipal Ta-Tung Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsu WL, Lu JH, Noda M, Wu CY, Liu JD, Sakakibara M, Tsai MH, Yu HS, Lin MW, Huang YB, Yan SJ, Yoshioka T. Derinat Protects Skin against Ultraviolet-B (UVB)-Induced Cellular Damage. Molecules. 2015 Nov 12;20(11):20297-311. doi: 10.3390/molecules201119693. PMID 26569211